CLINICAL TRIAL: NCT00971815
Title: Effects of 3 Months of SSRI-Treatment on Metabolism and HPA-axis in Young Men Born With Low Birth Weight - a Randomized, Double Blinded and Placebo-controlled Trial
Brief Title: Effects of 3 Months of Selective Serotonin Reuptake Inhibitor (SSRI)-Treatment on Metabolism and Hypothalamic-pituitary-adrenal (HPA)-Axis in Young Men Born With Low Birth Weight
Acronym: LBW-SSRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: M-20080132
Record Dates: First submitted 2009-06-02; First posted 2009-09-04 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2013-05

CONDITIONS: Insulin Resistance; Low Birth Weight; Type 2 Diabetes; Cardiovascular Disease; Melancholic Depression; Anxiety Disorders
Keywords: HPA-axis; fetal programming
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Depressive Disorder; Anxiety Disorders | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- escitalopram (Active Comparator): A pill containing Escitalopram
  Interventions: Drug: Escitalopram
- placebo (Placebo Comparator): a placebo pill
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Escitalopram — first week: 10mg/day. Then, treatment with 20mg/day is continued throughout a 3 months period of time.
  Other Names: Escitalopram (Cipralex)(H. Lundbeck A/S)
  Arms: escitalopram
Drug: placebo — 1/2 pill pr day first week, then 1 pill pr. day throughout a 3 months treatment period (90-118 ± 7days)
  Other Names: no other names
  Arms: placebo

SUMMARY:
Chronic stress has been proposed to be involved the development of western life-style diseases such as cardiovascular disease and type 2 diabetes (T2DM). At the same time chronic stress is also believed to cause psychiatric disease such as melancholic depression (MD)and anxiety disorders.

Accordingly, humans born with low birth weight (LBW) (ei. less than 5,0 LB) display an increased risk for T2DM and MD. Studies suggest stress and adrenal stress hormones (glucocorticoids) (GCC) might be involved in the development of both of these conditions.

Recent studies of animals born LBW suggest, that SSRI-compounds, usually employed in the treatment of MD-related diseases, reduces stress-responses and levels of stress hormones such adrenal steroids and at the same time has a positive influence on glucose metabolism.

In present study, the investigators aim to measure levels of GCC and stress and assess glucose metabolism in healthy young men (20-35 years) born LBW (40 subjects). The volume and structure of a certain brain area (ie. hippocampus) involved in regulation of adrenal GCC and known to be malfunctioning in chronically stressed individuals will be assessed by magnetic resonance imaging (MRI). Further metabolic examination will be accompanied by MRI spectroscopy of liver and muscle fat content as well as total fat content (Dexa-scanning) and contents of fat in the abdomen (by MRI) . Psychiatric well-ness and symptoms will be characterized by well-established questionnaires such as MDI and SCL-92 and responses as regards blood pressure, heart rate and changes in basal plasma concentrations of GCC and Epinephrine will be assessed while performing a Stroop Stress Test. Finally, a 24 hour blood pressure profile test will be included.

After this extensive examination program, subjects will be randomized to 3-4 months of treatment with either Escitalopram (an SSRI-compound) or Placebo. Subsequently, at the end of the treatment, the whole examination program will be repeated to detect potential beneficial changes.

A group of young normal birth weight men (20 subjects) will serve as a healthy baseline group for comparison and will not be exposed to any medical treatment.

This trial will add understanding to the mechanism underlying the development of type 2 diabetes and depression in LBW. Additionally, present trial might be capable of proposing a novel treatment strategy to prevent the development of these diseases in LBW man.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men 20-35 years old.
2. birth weight <2500g.
3. Born at gestational week 38- 40 (42).

Exclusion Criteria:

1. Diabetes, insulin-resistance or precursors in first degree relatives or maternal gestational diabetes.
2. Small parents(mother <160cm and/or father <170cm).
3. History of abuse of alcohol, medicine og drugs in the mother during pregnancy.
4. Liver of renal failure : s-ALAT > 2.5 normal upper limit (>175μM) or s-creatinine >125 μmol/l.
5. Co-morbidity that after at medical examination is considered to be a problem.
6. BMI>25.5
7. Smoking that is considered to be an issue as regards completing the study.
8. Treatment with a MAO-inhibitor.
9. Born before gestational week 38.
10. Participation in larger X-ray examinations such CT-scans during the last 12 months.
11. Participation in medical experiments or treatments involving intravenous administration of radioactive substances during the last
12. Ongoing medical treatment that will be considered a issue for completing the study.
13. Allergy towards the substance Escitalopram.
14. Metal parts in the body that contra-indicates MRI.
15. Ongoing medical treatment thrombocyte inhibiting substances such as NSAIDS.
16. Previous gastrointestinal bleeding or gastro-duodenal ulcers.
17. Depression during examination or treatment

16/05-2011: Criterias updated - added 17 and adjusted 6. from BMI >25 to BMI >25.5

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2011-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Changes in rate of glucose dissappearance | Changes in LBW-subjects from baseline vs. post-treatment after 3 months treatment with placebo or Escitalopram
Changes in the 24-hour AUC of free plasma cortisol | Changes in LBW-subjects from baseline vs. post-treatment after 3 months treatment with placebo or Escitalopram

SECONDARY OUTCOMES:
24 hour basal plasma cortisol/ACTH profile as measured every 3rd hour. | before and after 3 months of treatment with placebo or Escitalopram
hippocampic volume and structure as assessed by MRI | before and after 3 months of treatment with placebo or Escitalopram
  All limbic structures (amygdala, thalamus, hippocampus and ventromedial prefrontal cortex) were morphologically and volumetrically analyzed.
24 hour bloodpressure profile | before and after 3 months of treatment with placebo or Escitalopram
MRI spectroscopy of fat in skeletal muscle tissue | Before and after 3 months of treatment with placebo or Escitalopram
MRI spectroscopy of fat in liver | Before and after 3 months of treatment with placebo or Escitalopram
Abdominal fat as assessed by MRI | Before and after 3 months of treatment with placebo or Escitalopram
MDI questionnaire scores | Before and after 3 months of treatment with placebo or Escitalopram
SCL-92 questionnaire scores | Before and after 3 months of treatment with placebo or Escitalopram
Fasting blood lipid profile | Before and after 3 months of treatment with placebo or Escitalopram
Ratio between insulin and glucose concentrations in blood during an oral glucose tolerance test (OGTT) | Before and after 3 months of treatment with placebo or Escitalopram
Whole body fat content as assessed by a dexa scanning | Before and after 3 months of treatment with placebo or Escitalopram
Hepatic insulin sensitivity as assessed suppression of endogenous glucose production (calculated by infusion of 3H-labelled glucose) | Before and after 3 months of treatment with placebo or Escitalopram
10 pm to midnight basal plasma ACTH/cortisol concentration ratio as measured by blood sampling every 10th minute. | Before and after 3 months of treatment with placebo or Escitalopram
increase in blood pressure and heart rate during Stroops Stress test | Before and after 3 months of treatment with placebo or Escitalopram
Increase in plasma ACTH, cortisol and epinephrine concentrations during Stroops Stress Test | before and after 3 months of treatment with placebo or Escitalopram
SRPAS questionnaire scores | Before and after 3 months of treatment with placebo or Escitalopram
  Self Reported Physical Activity Questionaire
Actigraph GT3X activity monitoring | Before and after 3 months of treatment with placebo or Escitalopram
  Objective measurements of physical activity in 96 hours at home
Whole body bone mass density and T-/Z-scores as assessed by a dexa scanning | Before and after 3 months of treatment with placebo or Escitalopram
Plasma-Inflammation markers | Before and after 3 months of treatment with placebo or Escitalopram

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Dep M, Diabetes and Endocrinology Aarhus University Hospital, Aarhus Sygehus, Aarhus, Denmark

REFERENCES:
- [Derived] Buhl CS, Stodkilde-Jorgensen H, Videbech P, Vaag A, Moller N, Lund S, Buhl ES. Escitalopram Ameliorates Hypercortisolemia and Insulin Resistance in Low Birth Weight Men With Limbic Brain Alterations. J Clin Endocrinol Metab. 2018 Jan 1;103(1):115-124. doi: 10.1210/jc.2017-01438. PMID 29053851